CLINICAL TRIAL: NCT06301646
Title: A Randomized Controlled Trial To Explore the Effect of Oral vs. Nasal Enteral Nutrition Tube Feeding on Stroke Survivors in Social Interaction and Psychological Status
Brief Title: Oral Enteral Nutrition Tube Feeding on Stroke Survivors
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmadu Bello University Teaching Hospital (Other)
Responsible Party: Principal Investigator, Muhammad, Research Director, Ahmadu Bello University Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IOE-psy
Record Dates: First submitted 2024-03-04; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Cerebrovascular Accident
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- comprehensive rehabilitation therapy+Intermittent Oro-esophageal Tube Feeding (Experimental): Study lasts 15 days for each patient. The patients were given comprehensive rehabilitation therapy. The experimental group was provided the support of enteral nutrition by Intermittent Oro-esophageal Tube Feeding.
  Interventions: Device: Intermittent Oro-esophageal Tube Feeding; Behavioral: comprehensive rehabilitation therapy
- comprehensive rehabilitation therapy+Nasogastric Tube Feeding (Active Comparator): Study lasts 15 days for each patient. The patients were given comprehensive rehabilitation. The control group was provided the support of enteral nutrition by Nasogastric Tube Feeding.
  Interventions: Device: Nasogastric Tube Feeding; Behavioral: comprehensive rehabilitation therapy

INTERVENTIONS:
Device: Intermittent Oro-esophageal Tube Feeding — The specific procedure was as follows: the infant was placed in a semi-recumbent or sitting position with the head fixed. Before each feeding, the infant's oral and nasal secretions were to be cleared. An intermittent oro-esophageal tube was appropriately lubricated with water on the head part. The professional medical staff held the tube and slowly inserted it through one side of the mouth into the upper part of the esophagus. The depth of insertion depended on the patient's age and height. After each feeding, the tube was immediately removed, and the patient was held upright for at least 30 minutes in case of reflux.
  Arms: comprehensive rehabilitation therapy+Intermittent Oro-esophageal Tube Feeding
Device: Nasogastric Tube Feeding — Nasogastric Tube Feeding were used for feeding to provide nutritional support. Each feeding was administered by a nurse using the infant's mother's breast milk through the tube. The amount of each feeding varied from 20 to 100 ml depending on the age of the infant, with feedings given every 2 to 3 hours, approximately 10 times per day. The duration of each feeding procedure ranged from 10 to 20 minutes. The total daily intake ranged from 200 to 1000 ml. Each tube was kept indwelling for 5 to 7 days. When the tube needed to be replaced, it was removed after the last feeding of a day and a new tube was to be inserted through the other nostril on the following morning to continue the nutritional support.
  Arms: comprehensive rehabilitation therapy+Nasogastric Tube Feeding
Behavioral: comprehensive rehabilitation therapy — Both groups were given comprehensive rehabilitation therapy. The main intervention measures included: 1) non-invasive ventilator treatment, generally at least once every night and typically not exceeding continuous daily usage.; 2) attention to feeding and sleeping positions, with a recommended sleeping position of lateral recumbent and the head of the bed raised by 20-30°; 3) swallowing function training, such as tongue muscle stretching training, assisted anterior jaw protrusion training, lemon ice stimulation to the soft palate, pharyngeal wall, etc., generally 5 days per week, twice per day, 5-20 minutes each time; 4) pulmonary ultrashort wave therapy, generally at least 2-3 times a week, and not more than once a day; 5) physical therapy, such as intensive training for gross motor functions including lifting the head, turning over, sitting, crawling, standing, etc., generally 3-5 days per week, 1-2 times per day, 5-20 min each time.

SUMMARY:
The goal of this clinical trial is to explore Clinical Effect of Intermittent Oro-esophageal Tube Feeding in Dysphagic Stroke Survivors. The main questions it aims to answer are:

Can Intermittent Oro-esophageal Tube Feeding improve psychological status in Dysphagic Stroke Survivors? Can Intermittent Oro-esophageal Tube Feeding improve social interaction in Dysphagic Stroke Survivors? Patients will be randomly allocated into the control group or the experimental group, all under rehabilitation treatment, the experimental group will be given Intermittent Oro-esophageal Tube Feeding as nutrition support and the control group will be given Nasogastric tube. The study lasts 15 days for each patient. Researchers will compare the Social Functioning Scale, Social Support Questionnaire, Patients Health Questionnaire-9, General Anxiety Disorder-7 to see if the Intermittent Oro-esophageal Tube Feeding can help improve the symptom.

DETAILED DESCRIPTION:
Stroke is happening increasingly more. The goal of this clinical trial is to explore Clinical Effect of Intermittent Oro-esophageal Tube Feeding in Dysphagic Stroke Survivors. The main questions it aims to answer are:

Can Intermittent Oro-esophageal Tube Feeding improve psychological status in Dysphagic Stroke Survivors? Can Intermittent Oro-esophageal Tube Feeding improve social interaction in Dysphagic Stroke Survivors? Patients will be randomly allocated into the control group or the experimental group, all under rehabilitation treatment, the experimental group will be given Intermittent Oro-esophageal Tube Feeding as nutrition support and the control group will be given Nasogastric tube. The study lasts 15 days for each patient. Researchers will compare the Social Functioning Scale, Social Support Questionnaire, Patients Health Questionnaire-9, General Anxiety Disorder-7 to see if the Intermittent Oro-esophageal Tube Feeding can help improve the symptom.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years;
* meeting the diagnostic criteria of stroke;
* any degree of dysphagia at admission;
* steady vital signs, without severe cognitive impairment or sensory aphasia.
* transferred out within three weeks of hospitalization in the neurology department.

Exclusion Criteria:

* complicated with other neurological diseases;
* damaged mucosa or incomplete structure in nasopharynx;
* tracheostomy tube plugged;
* unfeasible to the support of parenteral nutrition;
* simultaneously suffering from liver, kidney failure, tumors, or hematological diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Social Functioning Scale | day 1 and day 15
  The Social Functioning Scale includes multiple subscales, and the score range is generally 0-100. Higher scores indicate better social functioning, while lower scores indicate limited social functioning or problems.

SECONDARY OUTCOMES:
Social Support Questionnaire | day 1 and day 15
  Social Support Questionnaire's score range is generally 0-100. Generally, higher scores are better and indicate more social support.
Anxiety | day 1 and day 15
  The anxiety was assessed using the Generalized Anxiety Disorder-7, including items related to fear, worry, attention, etc. The total score ranged from 0 to 21, which was positively correlated with potential anxiety.
Depression | day 1 and day 15
  The depression was assessed using the Patient Health Questionnaire-9, with aspects including mood swings, optimism, sleep quality, appetite, etc. The total score ranged from 0 to 27, which was positively correlated with potential depression.

CONTACTS AND LOCATIONS:
Overall Officials: Nieto Luis, Master, Study Director — Site Coordinator of United Medical Group

IPD SHARING:
Plan to Share IPD: No